CLINICAL TRIAL: NCT01144533
Title: Comparative Analysis of Intra-articular Injection of Steroid and/or Sodium Hyaluronate in Adhesive Capsulitis: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Comparative Analysis of Intra-articular Injection of Steroid and/or Sodium Hyaluronate in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Assistant Professor, SMG-SNU Boramae Medical Center., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRM-10-01
Record Dates: First submitted 2010-06-08; First posted 2010-06-15 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Isotonic saline (Placebo Comparator)
  Interventions: Procedure: isotonic saline injection into the glenohumeral joint
- Steroid (Experimental)
  Interventions: Procedure: steroid injection into the glenohumeral joint
- Hyaluronate (Experimental)
  Interventions: Procedure: sodium hyaluronate injection into the glenohumeral joint
- Steroid + Hyaluronate (Experimental)
  Interventions: Procedure: steroid and hyaluronate injection into the glenohumeral joint

INTERVENTIONS:
Procedure: isotonic saline injection into the glenohumeral joint — * Total volume of injection drugs: 8ml
  * isotonic saline 4ml + telebrix(contrast media) 4ml
  * The number of injections : only once during the study period
  * Injection site : glenohumeral joint
  * Material : 22-gauze spinal needle
  * Anteroposterior, lateral, and axial arthrography after injection was performed to determine accuracy and patterns of the injection.
  Arms: Isotonic saline
Procedure: steroid injection into the glenohumeral joint — * Total volume of injection drugs: 8ml
  * triamcinolone(40mg)1ml + isotonic saline 3ml + telebrix(contrast media)4ml
  * The number of injections : only once during the study period
  * Injection Site : glenohumeral joint
  * Material : 22-gauze spinal needle
  * Anteroposterior, lateral, and axial arthrography after injection was performed to determine accuracy and patterns of the injection.
  Arms: Steroid
Procedure: sodium hyaluronate injection into the glenohumeral joint — * Total volume of injection drugs: 8ml
  * sodium hyaluronate 2ml + isotonic saline 2ml + telebrix(contrast media)4ml
  * The number of injections : only once during the study period
  * Injection Site : glenohumeral joint
  * Material : 22-gauze spinal needle
  * Anteroposterior, lateral, and axial arthrography after injection was performed to determine accuracy and patterns of the injection.
  Arms: Hyaluronate
Procedure: steroid and hyaluronate injection into the glenohumeral joint — * Total volume of injection drugs: 8ml
  * triamcinolone(40mg)1ml + sodium hyaluronate 2ml + isotonic saline 1ml + telebrix(contrast media)4ml
  * The number of injections : only once during the study period
  * Injection Site : glenohumeral joint
  * Material : 22-gauze spinal needle
  * Anteroposterior, lateral, and axial arthrography after injection was performed to determine accuracy and patterns of the injection.
  Arms: Steroid + Hyaluronate

SUMMARY:
The purpose of this study is to compare the efficacy of intra-articular steroid injection, sodium hyaluronate injection, a combination of the two, and placebo in the treatment of adhesive capsulitis of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis : Adhesive Capsulitis of the Shoulder
* defining of adhesive capsulitis

  * the presence of shoulder pain
  * limitation of both active and passive movements of the glenohumeral joint of ≥25% in at list 2 directions(abduction,flexion,external rotation,internal rotation), as compared with the contralateral shoulder
* duration : symptomatic for < 1 year

Exclusion Criteria:

* bilateral symptoms
* uncontrolled diabetes mellitus
* overt hypothyroidism or hyperthyroidism
* previous shoulder surgery
* previous glenohumeral joint injection within recent 6months
* trauma to the shoulder the last six months that required hospital care
* neurological symptoms
* allergy to injection material
* secondary adhesive capsulitis
* systemic inflammatory ds including rheumatoid arthritis
* degenerative arthritis of shoulder joint
* infectious arthritis of shoulder joint
* dislocation of shoulder joint
* blood coagulation disease
* rotator cuff tear
* serious mental illness
* pregnancy
* fracture in shoulder lesion
* CVA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
SPADI Score (Shoulder Pain and Disability Index) | Postinjection 1month

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Jo, M.D., Ph.D, Principal Investigator — Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea